CLINICAL TRIAL: NCT06192836
Title: The Effect of Placental Removal Method and Uterine Massage at Cesarean Delivery on Preventing Postpartum Hemorrhage
Brief Title: Placental Removal Method And Uterine Massage On Preventing Postpartum Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Busra Lekesiz (Other Government)
Responsible Party: Sponsor-Investigator, Busra Lekesiz, Clinical Doctor, Ankara Etlik City Hospital
Organization: Ankara Etlik City Hospital (Other Government)
Other Study IDs: AEŞH-EK1-2023-562
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Postpartum Hemorrhage; Cesarean Section Complications; Uterine Atony
Keywords: Postpartum Atony; Uterine massage; Hemorrhage; Placenta; Cesarean
MeSH Terms: conditions — Postpartum Hemorrhage; Uterine Inertia; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group 1-: Operation will be performed by Dr BL
  1. Patients' postoperative 30th minute, 1st and 2nd hour systolic blood pressure, diastolic blood pressure, pulse rate, shock indexes
  2. Volume of diuresis at postoperative first six hours
  3. Hemoglobin and hematocrit values at preoperatively and 2nd, 6th, 24th hours postoperatively.
  4. Duration of the surgery.
  5. Need for additional dose of uterotonics
  6. Need for surgical methods to manage postpartum bleeding
  7. Duration of hospital stay
  Interventions: Procedure: Manual Removal 1
- Group 2: Operation will be performed by Dr AC
  1. Patients' postoperative 30th minute, 1st and 2nd hour systolic blood pressure, diastolic blood pressure, pulse rate, shock indexes
  2. Volume of diuresis at postoperative first six hours
  3. Hemoglobin and hematocrit values at preoperatively and 2nd, 6th, 24th hours postoperatively.
  4. Duration of the surgery.
  5. Need for additional dose of uterotonics
  6. Need for surgical methods to manage postpartum bleeding
  7. Duration of hospital stay
  Interventions: Procedure: Manual Removal 2
- Group 3: Operation will be performed by Dr SM
  1. Patients' postoperative 30th minute, 1st and 2nd hour systolic blood pressure, diastolic blood pressure, pulse rate, shock indexes
  2. Volume of diuresis at postoperative first six hours
  3. Hemoglobin and hematocrit values at preoperatively and 2nd, 6th, 24th hours postoperatively.
  4. Duration of the surgery.
  5. Need for additional dose of uterotonics
  6. Need for surgical methods to manage postpartum bleeding
  7. Duration of hospital stay
  Interventions: Procedure: Controlled Cord Traction 1
- Group 4: Operation will be performed by Dr AS
  1. Patients' postoperative 30th minute, 1st and 2nd hour systolic blood pressure, diastolic blood pressure, pulse rate, shock indexes
  2. Volume of diuresis at postoperative first six hours
  3. Hemoglobin and hematocrit values at preoperatively and 2nd, 6th, 24th hours postoperatively.
  4. Duration of the surgery.
  5. Need for additional dose of uterotonics
  6. Need for surgical methods to manage postpartum bleeding
  7. Duration of hospital stay
  Interventions: Procedure: Controlled Cord Traction 2
- Group 5: Operation will be performed by Dr EDD
  1. Patients' postoperative 30th minute, 1st and 2nd hour systolic blood pressure, diastolic blood pressure, pulse rate, shock indexes
  2. Volume of diuresis at postoperative first six hours
  3. Hemoglobin and hematocrit values at preoperatively and 2nd, 6th, 24th hours postoperatively.
  4. Duration of the surgery.
  5. Need for additional dose of uterotonics
  6. Need for surgical methods to manage postpartum bleeding
  7. Duration of hospital stay
  Interventions: Procedure: Controlled Cord Traction+Uterine Massage 1
- Group 6: Operation will be performed by Dr SKE
  1. Patients' postoperative 30th minute, 1st and 2nd hour systolic blood pressure, diastolic blood pressure, pulse rate, shock indexes
  2. Volume of diuresis at postoperative first six hours
  3. Hemoglobin and hematocrit values at preoperatively and 2nd, 6th, 24th hours postoperatively.
  4. Duration of the surgery.
  5. Need for additional dose of uterotonics
  6. Need for surgical methods to manage postpartum bleeding
  7. Duration of hospital stay
  Interventions: Procedure: Controlled Cord Traction+Uterine Massage 2

INTERVENTIONS:
Procedure: Manual Removal 1 — 1. Placenta will be removed manually
  2. Uterine incision will be repaired as double layered
  3. No uterine massage will be performed
  Groups: Group 1-
Procedure: Manual Removal 2 — 1. Placenta will be removed manually
  2. Uterine incision will be repaired as double layered
  3. Uterine massage will be performed for one minute duration, after uterine incision is closed
  Groups: Group 2
Procedure: Controlled Cord Traction 1 — 1. Placenta will be delivered via controlled cord traction
  2. Uterine incision will be repaired as double layered
  3. No uterine massage will be performed
  Groups: Group 3
Procedure: Controlled Cord Traction 2 — 1. Placenta will be delivered via controlled cord traction
  2. Uterine incision will be repaired as double layered
  3. Uterine massage will be performed for one minute duration, after uterine incision is closed
  Groups: Group 4
Procedure: Controlled Cord Traction+Uterine Massage 1 — 1. Placenta will be delivered via controlled cord traction plus uterine massage
  2. Uterine incision will be repaired as double layered
  3. No uterine massage will be performed after placental delivery
  Groups: Group 5
Procedure: Controlled Cord Traction+Uterine Massage 2 — 1. Placenta will be delivered via controlled cord traction plus uterine massage
  2. Uterine incision will be repaired as double layered
  3. Additional uterine massage for one minute duration will be performed after uterine incision is closed
  Groups: Group 6

SUMMARY:
Postpartum hemorrhage is the leading cause of maternal deaths in all over the world, especially in developing and underdeveloped countries. Medical and surgical methods exist for management of bleeding.

There are two surgical techniques for removal of the placenta on cesarean delivery, which are called manual removal and controlled cord traction. In manual removal group, the duration of surgery time might be shorter theoretically. Nevertheless, there are studies showing that manual removal of the placenta may increase postpartum endometritis and postpartum hemorrhage. The optimal method for removal of the placenta during the cesarean delivery remains uncertain (1).

It is a known fact that uterine massage after vaginal birth lowers the risk of postpartum hemorrhage (2) However, there is no study on how effective uterine massage is during cesarean delivery. In 2018, Saccone and colleagues wanted to publish a meta-analysis on the role of uterine massage in reducing postpartum bleeding during cesarean delivery, but when they examined the literature on the subject, they could not find a study which included only the group that gave birth by cesarean section and was free from bias. In the same publication, it was mentioned that it was necessary to investigate the effectiveness of uterine massage, which is a cost-free method that can reduce maternal morbidity in underdeveloped countries where maternal deaths due to postpartum bleeding are high, in cesarean section. (3)

DETAILED DESCRIPTION:
In this study, data of patients who underwent emergency cesarean delivery in the Department of Obstetrics and Gynecology, Ankara Etlik City Hospital, will be collected

The parameters to be examined in the research are as follows:

1. Patients' postoperative 30th minute, 1st and 2nd hour systolic blood pressure, diastolic blood pressure, pulse rate, shock indexes
2. Volume of diuresis at postoperative first six hours
3. Hemoglobin and hematocrit values at preoperatively and 2nd, 6th, 24th hours postoperatively.
4. Duration of the surgery.
5. Need for additional dose of uterotonics
6. Need for surgical methods to manage postpartum bleeding
7. Duration of hospital stay

The sample size of this study was calculated with the Gpower3.1 computer program.

The total number of samples with 90% power and 95% confidence interval was calculated as 338 patients. The number of volunteers to participate in our study is planned to be 360 in total, 60 volunteers for each group, across 6 groups. Results will be considered statistically significant for p< 0,05.

ELIGIBILITY:
Inclusion Criteria:

* Live singleton pregnancy of 37 0/7 weeks or more
* Without history of previous uterine atony
* No comorbidities
* No gestational hypertension or gestational diabetes mellitus

Exclusion Criteria:

* In utero fetal death
* Multiple gestation
* History of uterine atony
* Vaginal birth
* Previous history of cesarean delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: In our study, data of patients who underwent emergency cesarean delivery at the Department of Obstetrics and Gynecology, Ankara Etlik City Hospital, will be collected prospectively
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2024-01-10 (Estimated); Primary Completion 2024-12-22 (Estimated); Study Completion 2025-02-22 (Estimated)

PRIMARY OUTCOMES:
Comparison of patients' preoperative and postoperative hemoglobin levels | 24 hours
  The basal hemoglobin levels ( gr/dL) of the patients will be compared with the hemoglobin levels at 2nd, 6th and 24th hours.
Comparison of patients' preoperative and postoperative hematocrit levels | 24 hours
  The basal hematocrit levels (%) of the patients will be compared with the hematocrit levels at 2nd, 6th and 24th hours
Comparison of patients' postoperative shock indexes | 2 hours
  Postoperative 30th minute, 1st and 2nd hour shock indices (heart rate (beats per minute) / systolic blood pressure(mmHg) ) will be compared

SECONDARY OUTCOMES:
Comparison of the patients' postoperative heart rate | 2 hours
  Patients postoperative 30th minute, 1st and 2nd hour heart rate (beats in minute) will be compared
Comparison of the patients' postoperative systolic and diastolic blood pressure | 2 hours
  Patients postoperative 30th minute, 1st and 2nd hour systolic and diastolic blood pressure (mmHg) will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Busra Lekesiz, Principal Investigator — Ankara Etlik City Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anorlu RI, Maholwana B, Hofmeyr GJ. Methods of delivering the placenta at caesarean section. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD004737. doi: 10.1002/14651858.CD004737.pub2. PMID 18646109
- [Background] Hofmeyr GJ, Abdel-Aleem H, Abdel-Aleem MA. Uterine massage for preventing postpartum haemorrhage. Cochrane Database Syst Rev. 2013 Jul 1;2013(7):CD006431. doi: 10.1002/14651858.CD006431.pub3. PMID 23818022
- [Background] Saccone G, Caissutti C, Ciardulli A, Berghella V. Uterine massage for preventing postpartum hemorrhage at cesarean delivery: Which evidence? Eur J Obstet Gynecol Reprod Biol. 2018 Apr;223:64-67. doi: 10.1016/j.ejogrb.2018.02.023. Epub 2018 Feb 23. PMID 29499526